CLINICAL TRIAL: NCT07295873
Title: A Single-Center, Open-Label, Single-Arm, Self-Controlled Phase I Clinical Study to Evaluate Drug-Drug Interactions of Hydronidone With Entecavir, Tenofovir Disoproxil Fumarate, Tenofovir Alafenamide, and Tenofovir Amibufenamide in Healthy Chinese Subjects
Brief Title: Drug-Drug Interaction Study Between Hydronidone and Entecavir, Tenofovir Disoproxil Fumarate, Tenofovir Alafenamide, and Tenofovir Amibufenamide
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDN-F351-202505
Record Dates: First submitted 2025-12-10; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis B Liver Fibrosis; DDI (Drug-Drug Interaction)
Keywords: Hydronidone; F351
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Queue 1: Drug-Drug Interaction Study of Hydronidone Capsules and Entecavir (Experimental): Within each cohort, the study flow for enrolled subjects comprises three dosing periods: Period 1 consists of hydronidone capsules administered alone for 5 consecutive days; Period 2 consists of the chronic hepatitis B antiviral agent administered alone for 7 or 10 consecutive days; and Period 3 consists of concomitant administration of hydronidone capsules and the antiviral agent for 5 consecutive days. Subjects may be discharged from the study upon completion of the safety follow-up.
  hydronidone capsules,90 mg three times daily, under fasting conditions
  Interventions: Drug: Entecavir
- Queue 2: Drug-Drug Interaction Study of honyinone capsules and Tenofovir Disoproxil Fumarate; (Experimental): Within each cohort, the study flow for enrolled subjects comprises three dosing periods: Period 1 consists of hydronidone capsules administered alone for 5 consecutive days; Period 2 consists of the chronic hepatitis B antiviral agent administered alone for 7 or 10 consecutive days; and Period 3 consists of concomitant administration of hydronidone capsules and the antiviral agent for 5 consecutive days. Subjects may be discharged from the study upon completion of the safety follow-up.
  hydronidone capsules,90 mg three times daily, under fasting conditions
  Interventions: Drug: Tenofovir Disoproxil Fumarate（TDF）
- Drug-Drug Interaction Study of Fuzuloprim Capsules with Tenofovir Alafenamide (Experimental): Within each cohort, the study flow for enrolled subjects comprises three dosing periods: Period 1 consists of hydronidone capsules administered alone for 5 consecutive days; Period 2 consists of the chronic hepatitis B antiviral agent administered alone for 7 or 10 consecutive days; and Period 3 consists of concomitant administration of hydronidone capsules and the antiviral agent for 5 consecutive days. Subjects may be discharged from the study upon completion of the safety follow-up.
  hydronidone capsules,90 mg three times daily, under fasting conditions.
  Interventions: Drug: Tenofovir alafenamide（TAF）
- Queue 4: Drug-Drug Interaction Study of Hydronidone Capsules and Tenofovir Amibufenamide (Experimental): Within each cohort, the study flow for enrolled subjects comprises three dosing periods: Period 1 consists of hydronidone capsules administered alone for 5 consecutive days; Period 2 consists of the chronic hepatitis B antiviral agent administered alone for 7 or 10 consecutive days; and Period 3 consists of concomitant administration of hydronidone capsules and the antiviral agent for 5 consecutive days. Subjects may be discharged from the study upon completion of the safety follow-up.
  hydronidone capsules,90 mg three times daily, under fasting conditions.
  Interventions: Drug: Tenofovir Amibufenamide(TMF)

INTERVENTIONS:
Drug: Entecavir — 0.5 mg, taken orally on an empty stomach, once a day
  Arms: Queue 1: Drug-Drug Interaction Study of Hydronidone Capsules and Entecavir
Drug: Tenofovir Disoproxil Fumarate（TDF） — 300 mg, taken orally on an empty stomach, once a day
  Arms: Queue 2: Drug-Drug Interaction Study of honyinone capsules and Tenofovir Disoproxil Fumarate;
Drug: Tenofovir alafenamide（TAF） — 25 mg, single oral dose, under fasting conditions
  Arms: Drug-Drug Interaction Study of Fuzuloprim Capsules with Tenofovir Alafenamide
Drug: Tenofovir Amibufenamide(TMF) — 25 mg, single oral dose, under fasting conditions
  Arms: Queue 4: Drug-Drug Interaction Study of Hydronidone Capsules and Tenofovir Amibufenamide

SUMMARY:
The proposed indication for Hydronidone Capsules is chronic hepatitis B-associated liver fibrosis, which in clinical practice typically requires concomitant use with antiviral agents for chronic hepatitis B. The commonly used chronic hepatitis B antiviral agents include Entecavir, Tenofovir Disoproxil Fumarate (TDF), Tenofovir Alafenamide (TAF), and Tenofovir Amibufenamide (TMF).

This study aims to evaluate the drug-drug interaction (DDI) of Hydronidone Capsules 90 mg with Entecavir, Tenofovir Disoproxil Fumarate (TDF), Tenofovir Alafenamide (TAF), and Tenofovir Amibufenamide (TMF) respectively in healthy participants, to inform the preparation of post-marketing labeling and the development of concomitant dosing regimens in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Be fully informed about the trial and demonstrate understanding of its content, procedures, and potential adverse events related to the investigational product; voluntarily provide written informed consent; and be able to comply with all study procedures and complete the study in accordance with the protocol requirements.
* Male or female subjects aged 18 to 50 years, inclusive, at the time of signing informed consent.
* At screening, male subjects must weigh ≥50.0 kg and female subjects must weigh ≥45.0 kg, with a body mass index (BMI) between 19.0 and 26.0 kg/m², inclusive.
* At screening, all laboratory tests and related examinations (including vital signs, physical examination, 12-lead ECG, chest X-ray [PA view], abdominal ultrasound, etc.) must be within normal range or, if abnormal, determined by the investigator to be not clinically significant.

Exclusion Criteria:

* Presence of any clinically significant disease or medical history that, in the opinion of the investigator, may interfere with protocol compliance or completion of the study, including but not limited to abnormalities of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematologic system, immune system, psychiatric system, or endocrine/metabolic system.
* Positive results for any infectious disease screening tests at screening, including hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), human immunodeficiency virus antigen/antibody (HIV Ag/Ab), or Treponema pallidum antibody (TP Ab).
* History of drug or food allergies, or known hypersensitivity to the active pharmaceutical ingredients of the investigational medicinal products (hydronidone, entecavir, tenofovir disoproxil fumarate, tenofovir alafenamide, tenofovir amibufenamide) or to any of their excipients.
* Participants with rare genetic disorders of galactose intolerance, lactase deficiency, or glucose-galactose malabsorption;
* Subjects who have experienced a clinically significant major illness within 3 months prior to screening, or have undergone surgery affecting drug absorption, distribution, metabolism, or excretion (such as gastrointestinal, hepatic, or renal surgery) or other major surgery within this period, or plan to undergo surgery during the study;
* Subjects who have donated blood or experienced blood loss ≥400 mL within 3 months prior to dosing, or received blood transfusion or blood products within 4 weeks prior to dosing, or plan to donate blood during the study period;
* Subjects who have participated as a participant in any clinical trial and received investigational drug or device treatment within 3 months prior to dosing;
* Subjects who have taken any prescription medication, over-the-counter medication, vitamin products, or herbal medicines within 14 days or 5 half-lives (if known) prior to dosing, whichever is longer; or who have taken strong inhibitors or inducers of CYP3A4, P-glycoprotein (P-gp), breast cancer resistance protein (BCRP), OATP1B1, OATP1B3, or OAT1/3 within 4 weeks prior to screening; or any drugs known to cause QT/QTc interval prolongation or with a known risk of causing torsades de pointes (TdP) (see Appendix 2); or plan to use any chemical drugs, biological products, traditional Chinese medicines, or natural medicines that the investigator deems inappropriate during the trial period;
* Subjects who received vaccination within 4 weeks prior to screening, or plan to receive vaccination during the study period up to 1 month after the last dose; Subjects with a history of drug abuse within the past 5 years, or who used illicit drugs within 3 months prior to screening, or with a positive urine drug abuse screen at baseline;
* Subjects who regularly consumed alcohol within 6 months prior to dosing, i.e., more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol spirits or 150 mL of wine), or who refuse to abstain from alcohol or alcohol-containing products during the trial, or with a positive alcohol breath test at baseline;
* Subjects who smoked more than 5 cigarettes daily within 3 months prior to dosing, or who are unable to discontinue use of tobacco products during the trial period;
* Subjects with a history of blood-needle phobia/syncope, or unable to tolerate venous indwelling needle puncture;
* Subjects with special dietary requirements who cannot follow the standardized diet, or with difficulty swallowing;
* Subjects unable to avoid specific foods/diet during the trial period, including dragon fruit, mango, grapefruit or grapefruit-related citrus fruits (e.g., Seville orange, pomelo), star fruit, papaya, pomegranate or products thereof, and/or xanthine-containing diet, caffeine-containing food or beverages, strong tea, etc.;
* Subjects who consumed grapefruit or grapefruit-related citrus fruits (e.g., Seville orange, pomelo) or products thereof within 2 weeks prior to dosing, or who consumed specific diet (including dragon fruit, mango and/or xanthine-containing diet, caffeine-containing food or beverages, strong tea, etc.) within 48 hours prior to dosing, or engaged in strenuous exercise, or have other factors that may affect drug absorption, distribution, metabolism, or excretion;
* Pregnant or lactating women, or female subjects of childbearing potential with a positive serum pregnancy test at screening;
* Subjects of childbearing potential who do not agree to use effective contraceptive methods from the time of signing informed consent until 3 months after study completion (see Appendix 3), or do not agree to avoid freezing or donating eggs or sperm during this period;
* Subjects who, in the opinion of the investigator, have other reasons that render them unsuitable for participation in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma hydronidone PK parameters of hydronidone capsules : steady-state peak concentration (Cmax,ss); | 23 days
Plasma hydronidone PK parametersof hydronidone capsules : Area under the plasma concentration-time curve from time zero to 24 hours at steady state (AUC0-24h,ss) | 23 days
Primary PK parameters of plasma of entecavir : AUC0-24h,ss. | 23 days
Primary PK parameters of plasma of entecavir : Cmax,ss . | 23 days
Primary PK parameters of plasma tenofovir alafenamide (TAF) : AUC0-24h,ss. | 23 days
Primary PK parameters of plasma tenofovir alafenamide (TAF) : Cmax,ss . | 23 days
Primary PK parameters of tenofovir disoproxil fumarate tablets (TDF): Cmax,ss . | 20 days
Primary PK parameters of tenofovir disoproxil fumarate tablets (TDF): AUC0-24h,ss. | 20 days
Primary PK parameters of plasma tenofovir amibufenamide (TMF) : Cmax,ss . | 23 days
Primary PK parameters of plasma tenofovir amibufenamide (TMF) : AUC0-24h,ss. | 23 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Gaobo Hospital, Beijing, China